CLINICAL TRIAL: NCT03226184
Title: Sterilizing Effects of the Erbium:YAG Laser Upon Metal Implants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Lukas Kriechbaumer, MD, Medical University of Vienna
Other Study IDs: 2167/2013
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Orthopedic Devices Associated With Misadventures, Prosthetic and Other Implants, Materials and Accessory Devices
Keywords: Er:YAG laser, laser, biofilm removal, biofilm, disinfection, septic revision surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Even today, postoperative infection is the commonest complications after surgery although all aseptic precautions are taken and causes significant postoperative morbidity, mortality, prolongs hospital stay, and increases costs. Infections that are related to orthopaedic procedures are considered particularly severe when implantation materials are used which further increases the risk of infection and holds the risk of biofilm formation. This is of particular concern since biofilm-mediated infections are difficult to diagnose and effective treatments are lacking. Therefore, new strategies for implant infection are currently being researched worldwide. In this study the relatively new approach for infection control by using an Er:YAG laser was adapted to an orthopaedic and traumatologic setting. This laser vaporizes all water containing cells in a very effective, precise and predictable manner and shows only a minimal thermal damage.

Methods:

For preliminary testing 42 steel pins and 42 plates were cultivated with cocultures for 2 weeks. The minimally necessary laser energy for biofilm removal was determined. We subsequently compared the effectiveness of biofilm removal with the Er:YAG laser and a cleansing of the metal implants with Octenidine soaked gauze. The temperature rise within the metal during the laser procedure was also measured.

In order to achieve an approximation to a clinical setting we want to compared the same effectiveness of biofilm removal similarly on steel pins directly after explantation from patients treated with external fixators for at least 2 weeks. Sonication and SEM will be used for analysis.

Preliminary Results Laser fluences exceeding 2.8J/cm2 caused a complete extinction of all living cells by a single laser impulse. Temperature rise within the implant is dependent on repetition frequency but overall negligible.

The effectiveness of biofilm removal after cleansing with Octenidine soaked gauze and irradiation with the Er:YAG laser will be evaluated on cultivated and extracted pins.

Conclusions We want to compare the effectiveness of the Er:YAG laser and Octenidine in the removal of biofilms from half-pins. We hypothesize that thee Er:YAG laser offers a secure, complete and non toxic removal of all kinds of pathogens from steel implants without damaging the implant or possible development of resistances. The precise non-contact removal of adjacent tissue could be an advantage over other disinfectants.

Level of Evidence (II-a)

Clinical Relevance:

Having one more arrow in the quiver for disinfection of percutaneous implants or for septic revision surgery when osteosynthesis equipment or arthroplasties are meant to be left in place would be extremely desirable.

ELIGIBILITY:
Inclusion Criteria:

All patients that are treated with external fixators for at least 2 weeks and patients whose implants have to be removed during septic revision surgery.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: same as inclusion criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Completeness of biofilm removal | 2 years
  Is the Er:YAG laser able to remova a microbial biofilm from cultivated or infected implants

SECONDARY OUTCOMES:
Side effects | 2 years
  Are there side effect to be expected from laser Irradiation either for the implant or for the surrounding tissue in a possible clinical setting

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Traumatology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No